CLINICAL TRIAL: NCT02654886
Title: Safety and Effectiveness of Resistance Exercise Training in Patients With Late Onset Pompe Disease- A Pilot Study
Brief Title: Safety and Effectiveness of Resistance Exercise Training in Patients With Pompe Disease.
Acronym: ExercisPompe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Virginia Kimonis, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS# 2013-9365
Record Dates: First submitted 2015-12-10; First posted 2016-01-13 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pompe Disease; Muscle Weakness
Keywords: exercise; Pompe disease; Pompe
MeSH Terms: conditions — Glycogen Storage Disease Type II; Muscle Weakness; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistance Exercise Training (Experimental): Participants will be given a regimen of resistance training after a 2 month observation period. Participants will be trained for 6 months (total= 72 training sessions). Two muscle groups (limbs) would be included in the resistance-training program. Participants will also be initiated with Respiratory muscle strength training using pressure-threshold respiratory trainers.
  Interventions: Other: Resistance Exercise Training

INTERVENTIONS:
Other: Resistance Exercise Training — Resistance Exercise Training: knee extension and elbow flexion each 3 times per week 3 sets each session; 10 reps/set for 6 months
  Respiratory muscle strength training: 25 repetitions -twice daily, 6 days/week for 6 months

SUMMARY:
The purpose of this research study is to determine if exercise will help improve muscle strength, endurance, and quality of life in individuals with Pompe disease. This is a research study to further define the outcome of patients with Pompe disease treated with a combined diet and exercise therapy.

DETAILED DESCRIPTION:
Eligibility: Subjects that are age 16 years or older, have been diagnosed with Pompe disease by genetic testing, and are showing symptoms such as muscle weakness

Time Commitment:

The study will last for 8 months. This study consists of a baseline visit of and return visits at week 9, week 16, week 24, and week 32. At the week 9 visit the subject will be given an individualized exercise plan which will be carried out over the next 24 weeks. The subject will be asked to return for three more visits at week16, week 24 and week 32. The 24 week training period will involve 3 workouts a week approximately 15-30 minutes each. It will also involve a breathing exercise that the subject can do at home twice daily for 10-15 minutes per session. The study visits will include the exercise plan, physical exam, blood draw and questionnaires.

Anticipated Benefits:

The possible benefits include a delay in progression of muscle weakness. The knowledge gained from this study will help researchers understand the effect of exercise on the disease. This may eventually lead to new forms of prevention of symptom onset in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Able to fully consent to the protocol.
2. Physically able to perform resistance exercises for 12 weeks.
3. Patients with a confirmed diagnosis of Pompe disease.
4. Age 16 years to 75 years.
5. Currently receiving ERT.
6. Patient on ERT for at least 1year.

Exclusion Criteria:

1. Patients with no confirmed diagnosis of Pompe disease, either by GAA enzyme deficiency from any tissue and/or molecular testing revealing two GAA gene mutations
2. Unable to walk or cycle
3. Unable to consent to the study/ procedures
4. Women who are pregnant or breastfeeding
5. Heart disease
6. Patients with any metal inside their body such as metallic clips used for vascular repairs and/or implanted devices such as cardiac pacemakers which would prevent them from doing the MRI.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Isometric muscle strength change from week 8 through week 32 | Eight months

SECONDARY OUTCOMES:
6 Minute Walk Test change from week 8 through week 32 | Eight months
Maximum Inspiratory Pressures percent change from week 8 through week 32 | Eight months
MRC score change from week 8 through week 32 | Eight months
Muscle volume and texture change from week 8 through week 32 using MR Imaging | Eight months
Glycogen content change in quadriceps muscle from week 8 through week 32 | Eight months
GAA enzyme activity change from week 8 through week 32 | Eight months
HEX4 change from week 8 through week 32 | Eight months
Other spirometry parameters change from week 8 through week 32 | Eight months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kimonis, MD MRCP, Principal Investigator — University of California, Irvine
Locations (1):
- UCI ICTS (Institute for Clinical and Translational Science), Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to partcipants after data is published in a peer reviewed journal.

REFERENCES:
- [Background] Bembi B, Pisa FE, Confalonieri M, Ciana G, Fiumara A, Parini R, Rigoldi M, Moglia A, Costa A, Carlucci A, Danesino C, Pittis MG, Dardis A, Ravaglia S. Long-term observational, non-randomized study of enzyme replacement therapy in late-onset glycogenosis type II. J Inherit Metab Dis. 2010 Dec;33(6):727-35. doi: 10.1007/s10545-010-9201-8. Epub 2010 Sep 14. PMID 20838899
- [Background] Bodamer OA, Leonard JV, Halliday D. Dietary treatment in late-onset acid maltase deficiency. Eur J Pediatr. 1997 Aug;156 Suppl 1:S39-42. doi: 10.1007/pl00014270. PMID 9266214
- [Background] Schoser B, Hill V, Raben N. Therapeutic approaches in glycogen storage disease type II/Pompe Disease. Neurotherapeutics. 2008 Oct;5(4):569-78. doi: 10.1016/j.nurt.2008.08.009. PMID 19019308
- [Background] Slonim AE, Coleman RA, McElligot MA, Najjar J, Hirschhorn K, Labadie GU, Mrak R, Evans OB, Shipp E, Presson R. Improvement of muscle function in acid maltase deficiency by high-protein therapy. Neurology. 1983 Jan;33(1):34-8. doi: 10.1212/wnl.33.1.34. PMID 6401355
- [Background] Slonim AE, Bulone L, Goldberg T, Minikes J, Slonim E, Galanko J, Martiniuk F. Modification of the natural history of adult-onset acid maltase deficiency by nutrition and exercise therapy. Muscle Nerve. 2007 Jan;35(1):70-7. doi: 10.1002/mus.20665. PMID 17022069
- [Background] Sveen ML, Jeppesen TD, Hauerslev S, Kober L, Krag TO, Vissing J. Endurance training improves fitness and strength in patients with Becker muscular dystrophy. Brain. 2008 Nov;131(Pt 11):2824-31. doi: 10.1093/brain/awn189. Epub 2008 Sep 6. PMID 18776212
- [Background] Terzis G, Dimopoulos F, Papadimas GK, Papadopoulos C, Spengos K, Fatouros I, Kavouras SA, Manta P. Effect of aerobic and resistance exercise training on late-onset Pompe disease patients receiving enzyme replacement therapy. Mol Genet Metab. 2011 Nov;104(3):279-83. doi: 10.1016/j.ymgme.2011.05.013. Epub 2011 May 19. PMID 21640624
- [Background] Winkel LP, Van den Hout JM, Kamphoven JH, Disseldorp JA, Remmerswaal M, Arts WF, Loonen MC, Vulto AG, Van Doorn PA, De Jong G, Hop W, Smit GP, Shapira SK, Boer MA, van Diggelen OP, Reuser AJ, Van der Ploeg AT. Enzyme replacement therapy in late-onset Pompe's disease: a three-year follow-up. Ann Neurol. 2004 Apr;55(4):495-502. doi: 10.1002/ana.20019. PMID 15048888
- [Background] Jones HN, Crisp KD, Robey RR, Case LE, Kravitz RM, Kishnani PS. Respiratory muscle training (RMT) in late-onset Pompe disease (LOPD): Effects of training and detraining. Mol Genet Metab. 2016 Feb;117(2):120-8. doi: 10.1016/j.ymgme.2015.09.003. Epub 2015 Sep 8. PMID 26381077
- [Background] van den Berg LE, Favejee MM, Wens SC, Kruijshaar ME, Praet SF, Reuser AJ, Bussmann JB, van Doorn PA, van der Ploeg AT. Safety and efficacy of exercise training in adults with Pompe disease: evalution of endurance, muscle strength and core stability before and after a 12 week training program. Orphanet J Rare Dis. 2015 Jul 19;10:87. doi: 10.1186/s13023-015-0303-0. PMID 26187632